CLINICAL TRIAL: NCT00057850
Title: Phase I/II Trial of the Epothilone B Analogue BMS 247550 (NSC 710428)/Cisplatin in Patients With Metastatic or Recurrent Squamous Cell Carcinoma of the Head and Neck
Brief Title: BMS-247550 Plus Cisplatin in Treating Patients With Metastatic or Recurrent Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02523; UPCC-04302; NCI-5787; CDR0000276716 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2003-04

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; salivary gland squamous cell carcinoma; stage IV salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — Cisplatin; ixabepilone

ARMS (1):
- Arm I (Experimental): Phase I: Patients receive BMS-247550 IV over 3 hours and cisplatin IV over 30-60 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of BMS-247550 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, up to 10 additional patients receive treatment as above at the recommended phase II dose of BMS-247550.
  Phase II: Patients receive treatment as in Phase I at the recommended phase II dose of BMS-247550.
  Interventions: Drug: cisplatin; Drug: ixabepilone

INTERVENTIONS:
Drug: cisplatin
Drug: ixabepilone

SUMMARY:
Phase I/II trial to study the effectiveness of combining BMS-247550 with cisplatin in treating patients who have metastatic or recurrent head and neck cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the recommended phase II dose of BMS-247550 when administered with cisplatin in patients with metastatic or recurrent squamous cell carcinoma of the head and neck. (Phase I) II. Determine the toxic effects of this regimen in these patients. III. Determine the response rate, time to progression, and survival of patients treated with this regimen. (Phase II) IV. Determine the pharmacokinetics of this regimen in these patients. V. Correlate selected markers from peripheral blood mononuclear cells and tumor samples with toxicity and response in patients treated with this regimen.

OUTLINE: This is an open-label, dose-escalation study of BMS-247550.

Phase I: Patients receive BMS-247550 IV over 3 hours and cisplatin IV over 30-60 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of BMS-247550 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, up to 10 additional patients receive treatment as above at the recommended phase II dose of BMS-247550.

Phase II: Patients receive treatment as in Phase I at the recommended phase II dose of BMS-247550.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the head and neck considered incurable by surgery or radiotherapy

  * No nasopharyngeal disease as primary site
* Extensive, local-regional or distant metastatic disease

  * Newly diagnosed OR
  * Recurrent disease after initial treatment with surgery or radiotherapy (including neoadjuvant chemotherapy or concurrent chemoradiotherapy)
* Measurable disease

  * If only site of measurable disease is in a previously irradiated area, disease progression after radiotherapy must be documented

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Hematopoietic

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 2.0 mg/dL
* Transaminases no greater than 2 times upper limit of normal (ULN) (5 times ULN if liver involvement)

Renal

* Creatinine no greater than 1.5 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No evidence of active infection
* No other malignancy within the past 2 years except curatively treated stage 0 or I cancer

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No prior chemotherapy for recurrent disease

Radiotherapy

* At least 6 months since prior radiotherapy and recovered

Surgery

* Recovered from prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2002-01; Primary Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane M. Hershock, MD, PhD, Study Chair — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States